CLINICAL TRIAL: NCT06706791
Title: Effect of Empagliflozin on Quality of Life in Chronic Heart Failure Patients With Diabetes Mellitus Type II
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Fazaia Ruth Pfau Medical College (Other)
Responsible Party: Principal Investigator, Tooba Riaz, clinical reseacher resident in FCPS Pharmacology, Fazaia Ruth Pfau Medical College
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FRPMC-IRB-2024-64; FMC,Air university (Other: Air university)
Record Dates: First submitted 2024-11-22; First posted 2024-11-27 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Chronic Heart Failure
Keywords: CHF DM type II
MeSH Terms: interventions — empagliflozin

STUDY DESIGN:
Intervention Model Description: This is a comparative clinical study with randomized groups. Participants will be allocated to either the Empagliflozin group or the placebo group alongside standard therapy.
  Blinding will be done by assigning drug to participants according to computer generated numbers in 2 groups in 1:1 ratio.
  Empagliflozin Group: taking Empagliflozin 10mg once daily per oral along with standard treatment. Their quality of life assessed by using Kansas City Cardiomyopathy questionnaire. Placebo Group: Identical placebo tablets, following the same dose and schedule as the Empagliflozin group along with standard treatment of chronic heart failure.
  Duration 18 months Setting Will take place in Fazaia Ruth Pfau medical college and hospital and NICVD hospital Karachi.
Who Masked: Participant, Investigator
Masking Description: The study will employ a double blind masking approach to ensure unbiased results and mainbtain the integrity of data participants masking; participants will be unaware of whether they are receiving Empagliflozin or placebo investigator masking; healthcare professionals and investigators administering the treatment will not know the treatment assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental arm, Palcebo controlled group (Experimental): Experimental arm, taking empagliflozin 10mg once daily along with standard treatment.
  Interventions: Drug: Empagliflozin 10 MG
- Palcebo controlled group (Placebo Comparator): Palcebo controlled group patient receiving placebo to compare with empagliflozin along with standard treatment.
  Interventions: Drug: Empagliflozin 10 MG

INTERVENTIONS:
Drug: Empagliflozin 10 MG — participants will be divided in two groups one group will empagliflozin 10mg once daily along with standard treatment secong group receiving placebo once daily along with standard treatment.
  Other Names: Horizon,

SUMMARY:
Effect of Empagliflozin on Quality of Life in patient of Chronic Heart Failure with Diabetes Mellitus Type II. As per ESC Guidelines Empagliflozin is recommended as part of the first-line treatment for HFrEF, irrespective of diabetes status.

As per American College of Cardiology (ACC)/American Heart Association (AHA) Empagliflozin is recommended in both diabetic and non-diabetic HF (especially beneficial in patients with HFrEF and HFpEF).

The aim of my study is to assess the impact of Empagliflozin on quality of life in Pakistani patients, considering the genetic, environmental and cultural factors.

The study will also explore whether Empagliflozin can offer cost-effective option for managing chronic heart failure and diabetes, potentially reducing the economic burden on both patients and health care system.

DETAILED DESCRIPTION:
Effect of Empagliflozin on Quality of Life in patient of Chronic Heart Failure with Diabetes Mellitus Type II. As per ESC Guidelines Empagliflozin is recommended as part of the first-line treatment for HFrEF, irrespective of diabetes status.

This is a comparative clinical study with randomized groups. Participants will be allocated to either the Empagliflozin group or the placebo group alongside standard therapy.

Blinding will be done by assigning drug to participants according to computer generated numbers in 2 groups in 1:1 ratio.

Empagliflozin Group: taking Empagliflozin 10mg once daily per oral along with standard treatment. Their quality of life assessed by using Kansas City Cardiomyopathy questionnaire. Placebo Group: Identical placebo tablets, following the same dose and schedule as the Empagliflozin group along with standard treatment of chronic heart failure.

Duration is of18 months. Will take place in Fazaia Ruth Pfau medical college and hospital and NICVD hospital Karachi.

ELIGIBILITY:
Inclusion Criteria:

1. Age 40-70 years at time of screening.
2. Both Men and women are included in study.
3. Patients with chronic heart failure and currently categorized in class II-IV heart failure as per NHYA classification having ejection fraction less than 40%.
4. Patients having NT- proBNP levels greater than 25pg/ml.
5. Diabetic patient diagnosed (HbA1c > 6.5mg/dl) and currently taking antidiabetic medicine.

Exclusion Criteria:

1. Pregnant female.
2. Patient with end stage renal disease (ESRD).
3. Patient with acute decompensated heart failure.
4. Acute coronary syndrome patients.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
improvement in Kansas city cardiomyopathy questionnaire scoring | 18 months
  Primary outcome measure will be the improvement in quality of life indicating by change in Kansas City cardiomyopathy questionnaire (KCCQ) scoring. higher value indicates better results.

SECONDARY OUTCOMES:
assessment of NT-pro-BNP levels. | 18 months
  Secondary outcome measures will include the change in NT-pro-BNP levels.lower values indicates better results

CONTACTS AND LOCATIONS:
Overall Officials: Tooba Riaz, MBBS, Principal Investigator — Fazaia Ruth Pfau Medical College
Locations (1):
- Fazaia Ruth Pfau Hospital, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No
it will be shared if required by relevent authorities

REFERENCES:
- [Background] McDonagh TA, Metra M, Adamo M, Gardner RS, Baumbach A, Bohm M, Burri H, Butler J, Celutkiene J, Chioncel O, Cleland JGF, Coats AJS, Crespo-Leiro MG, Farmakis D, Gilard M, Heymans S, Hoes AW, Jaarsma T, Jankowska EA, Lainscak M, Lam CSP, Lyon AR, McMurray JJV, Mebazaa A, Mindham R, Muneretto C, Francesco Piepoli M, Price S, Rosano GMC, Ruschitzka F, Kathrine Skibelund A; ESC Scientific Document Group. 2021 ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure. Eur Heart J. 2021 Sep 21;42(36):3599-3726. doi: 10.1093/eurheartj/ehab368. No abstract available. PMID 34447992
- [Background] Dunlay SM, Roger VL, Redfield MM. Epidemiology of heart failure with preserved ejection fraction. Nat Rev Cardiol. 2017 Oct;14(10):591-602. doi: 10.1038/nrcardio.2017.65. Epub 2017 May 11. PMID 28492288
- [Background] Januzzi JL Jr, Zannad F, Anker SD, Butler J, Filippatos G, Pocock SJ, Ferreira JP, Sattar N, Verma S, Vedin O, Schnee J, Iwata T, Cotton D, Packer M; EMPEROR-Reduced Trial Committees and Investigators. Prognostic Importance of NT-proBNP and Effect of Empagliflozin in the EMPEROR-Reduced Trial. J Am Coll Cardiol. 2021 Sep 28;78(13):1321-1332. doi: 10.1016/j.jacc.2021.07.046. PMID 34556318
- [Background] Januzzi JL Jr, Ahmad T, Mulder H, Coles A, Anstrom KJ, Adams KF, Ezekowitz JA, Fiuzat M, Houston-Miller N, Mark DB, Pina IL, Passmore G, Whellan DJ, Cooper LS, Leifer ES, Desvigne-Nickens P, Felker GM, O'Connor CM. Natriuretic Peptide Response and Outcomes in Chronic Heart Failure With Reduced Ejection Fraction. J Am Coll Cardiol. 2019 Sep 3;74(9):1205-1217. doi: 10.1016/j.jacc.2019.06.055. PMID 31466618
- [Result] Zinman B, Wanner C, Lachin JM, Fitchett D, Bluhmki E, Hantel S, Mattheus M, Devins T, Johansen OE, Woerle HJ, Broedl UC, Inzucchi SE; EMPA-REG OUTCOME Investigators. Empagliflozin, Cardiovascular Outcomes, and Mortality in Type 2 Diabetes. N Engl J Med. 2015 Nov 26;373(22):2117-28. doi: 10.1056/NEJMoa1504720. Epub 2015 Sep 17. PMID 26378978
- [Result] Heidenreich PA, Bozkurt B, Aguilar D, Allen LA, Byun JJ, Colvin MM, Deswal A, Drazner MH, Dunlay SM, Evers LR, Fang JC, Fedson SE, Fonarow GC, Hayek SS, Hernandez AF, Khazanie P, Kittleson MM, Lee CS, Link MS, Milano CA, Nnacheta LC, Sandhu AT, Stevenson LW, Vardeny O, Vest AR, Yancy CW. 2022 AHA/ACC/HFSA Guideline for the Management of Heart Failure: A Report of the American College of Cardiology/American Heart Association Joint Committee on Clinical Practice Guidelines. J Am Coll Cardiol. 2022 May 3;79(17):e263-e421. doi: 10.1016/j.jacc.2021.12.012. Epub 2022 Apr 1. PMID 35379503
- [Result] Packer M, Anker SD, Butler J, Filippatos G, Pocock SJ, Carson P, Januzzi J, Verma S, Tsutsui H, Brueckmann M, Jamal W, Kimura K, Schnee J, Zeller C, Cotton D, Bocchi E, Bohm M, Choi DJ, Chopra V, Chuquiure E, Giannetti N, Janssens S, Zhang J, Gonzalez Juanatey JR, Kaul S, Brunner-La Rocca HP, Merkely B, Nicholls SJ, Perrone S, Pina I, Ponikowski P, Sattar N, Senni M, Seronde MF, Spinar J, Squire I, Taddei S, Wanner C, Zannad F; EMPEROR-Reduced Trial Investigators. Cardiovascular and Renal Outcomes with Empagliflozin in Heart Failure. N Engl J Med. 2020 Oct 8;383(15):1413-1424. doi: 10.1056/NEJMoa2022190. Epub 2020 Aug 28. PMID 32865377
- [Result] Stubblefield WB, Jenkins CA, Liu D, Storrow AB, Spertus JA, Pang PS, Levy PD, Butler J, Chang AM, Char D, Diercks DB, Fermann GJ, Han JH, Hiestand BC, Hogan CJ, Khan Y, Lee S, Lindenfeld JM, McNaughton CD, Miller K, Peacock WF, Schrock JW, Self WH, Singer AJ, Sterling SA, Collins SP. Improvement in Kansas City Cardiomyopathy Questionnaire Scores After a Self-Care Intervention in Patients With Acute Heart Failure Discharged From the Emergency Department. Circ Cardiovasc Qual Outcomes. 2021 Oct;14(10):e007956. doi: 10.1161/CIRCOUTCOMES.121.007956. Epub 2021 Sep 24. PMID 34555929
- See also: pubmed — https://pubmed.ncbi.nlm.nih.gov/